CLINICAL TRIAL: NCT04574999
Title: Randomized, Double-blind, Placebo-controlled, Parallel Groups, Multicentre Study, to Determine Efficacy and Safety of a Low Concentration Estriol (ITFE-2026 0.005%) by Vaginal Route in the Treatment of Postmenopausal Vaginal Atrophy.
Brief Title: Study to Determine Efficacy & Safety of a Low Concentration Estriol (0.005%) in Postmenopausal Vaginal Atrophy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Italfarmaco S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITFE-2026C2
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Results first posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-09

CONDITIONS: Vaginal Atrophy
Keywords: Postmenopausal women
MeSH Terms: interventions — Estriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study drug, 0.005% Estriol vaginal gel, and its vehicle in gel (placebo) will have identical appearance, same aroma and the same texture in order to maintain the double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.005% Estriol group (Experimental): 0.005% Estriol (50 μg/g) gel for vaginal administration. Route: Vaginal by a cannula inserted deep inside the vagina Single dose: 1 g of gel Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: single application 2 times per week.
  Interventions: Drug: Estriol
- Placebo group (Placebo Comparator): Placebo gel for vaginal administration. Route: Vaginal by a cannula inserted deep inside the vagina Single dose: 1 g of gel Dosage schedule: Weeks 1-3: single daily application Weeks 4-12: single application 2 times per week.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Estriol — Gel for vaginal application
  Other Names: 16α-hydroxyestradiol or as estra-1,3,5(10)-triene-3,16α,17β-triol
  Arms: 0.005% Estriol group
Other: Placebo — Gel for vaginal application
  Arms: Placebo group

SUMMARY:
Randomized, double-blind, placebo-controlled multicentre study, with parallel groups, to determine the efficacy and safety of a new low-concentration estriol formulation (ITFE-2026 0.005%) for application by vaginal route in the treatment of postmenopausal vaginal atrophy.

Primary objective:

• To evaluate the efficacy of 0.005% Estriol vaginal gel by evaluation of the change in the maturation value of the vaginal epithelium (MV) after 12 weeks of treatment.

Secondary objectives:

* To determine the variation of the vaginal pH, as well as symptoms and signs suggestive of vaginal atrophy after 12 weeks of treatment.
* To study the variation of the MV, pH and symptoms and signs suggestive of vaginal atrophy after an initial observation period of 3 weeks.
* To evaluate the safety of 0.005% Estriol vaginal gel
* To evaluate the acceptability of 0.005% Estriol vaginal gel

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled multicentre study, with parallel groups, to determine the efficacy and safety of a new low-concentration estriol formulation (ITFE-2026 0.005%) for application by vaginal route in the treatment of postmenopausal vaginal atrophy.

Eligible patients were randomised in a ratio of 2:1 to 0.005% Estriol vaginal gel : placebo. Each patient was treated for 12 weeks followed by a one-month observational period. The patients attended the study centre at baseline and at 3, 8 and 12 weeks after start of treatment. Vaginal cytology was performed at baseline and at weeks 3 and 12; the vaginal pH and the signs and symptoms of vaginal atrophy were recorded at baseline and after 3 and 12 weeks of treatment. Vital signs, gynaecological exploration and changes in health and concomitant medication were documented at each visit. Transvaginal ultrasound was performed at screening and week 12. The investigators telephoned the patient approximately one month after the final visit to check if the patient had experienced any adverse events since the final visit. Two independent cytopathologists assessed the maturation value of each cytology sample at the end of the study.

ELIGIBILITY:
Main Inclusion Criteria:

* Women of any age.
* Menopause with amenorrhea time ≥ 2 years, either due to natural or surgical menopause (bilateral oophorectomy).
* Presence of symptoms and signs of atrophy of the vaginal mucosa including at minimum vaginal dryness as a symptom stated by the patient, together with at least one sign of the disease verified by the investigator.

  * As symptoms the patient could state vaginal dryness, pruritus, burning, dyspareunia, dysuria or any other symptom that the investigator considered related to the presence of vaginal atrophy.
  * As signs the investigator assessed in the gynaecological examination with a speculum, a thinned vaginal mucosa or with flattening of folds, a dry, fragile and pale vaginal mucosa, the presence of petechiae or any other sign that the investigator considered indicative of the existence of vaginal atrophy
* Patients with mammography carried out in the period of one year prior to inclusion in the study.
* Patients able to understand the nature and purpose of the study, to cooperate with the investigator and meet the study requirements.
* Patients who gave written informed consent to participate in the study.

Exclusion Criteria:

* Patients with contraindications for hormone therapy with estrogens because they had a history of:

  * Malignant or premalignant lesions of the breasts or endometrium.
  * Pathology of malignant colon tumour.
  * Malignant melanoma
  * Hepatic tumour pathology
  * Venous thromboembolic conditions (deep vein thrombosis, pulmonary embolism) or arterial thromboembolic conditions (angor pectoris, myocardial infarction, cerebrovascular accident), peripheral arterial disease, mesenteric artery thrombosis, renal artery thrombosis
  * Coagulopathies
  * Vaginal bleeding of unknown etiology
* Patients who had abnormal laboratory values at the start of the study that the investigator considered clinically relevant for the purposes of the present study.
* Patients with signs and symptoms suggestive of infection of the genital or urinary tract at the start of the study.
* Patients with any medical-surgical pathology, which was uncontrolled at the time of inclusion in the study.
* Patients with any acute process whose handling or evolution the investigator considered could interfere in the development of the study.
* Patients with endometrial thickness equal to or greater than 4 mm measured by transvaginal ultrasound.
* Patients with grade II or higher uterovaginal prolapse.
* Patients who had received any type of vulvovaginal treatment in the 15 days prior to the start of the study.
* Patients who had received phytoestrogens in the period of one month prior to the start of the study, including administration by vaginal route.
* Patients who had received hormone therapy in the period of 3 months prior to the start of the study, including the administration of estrogens by vaginal route.
* Patients on treatment with drugs described in section 7.3 of the protocol
* Patients with a history of allergy to any of the components of the medication under study (see the composition in section 3.3. of the protocol).
* Patients who had participated in the experimental evaluation of any drug during the 8 weeks before the start of the present study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2008-01-25 (Actual); Primary Completion 2009-02-23 (Actual); Study Completion 2009-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Ferrer Barriendos, MD, PhD, Principal Investigator — Hospital Universitario Central de Asturias
Locations (12):
- Spain (12):
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Hospital Ruber Internacional, Madrid, Castiglia
  - Centre Mèdic Teknon S.L., Barcelona, Catalonia
  - Fundació de Gestió Sanitària de l'Hospital de la Santa. Creu i Sant Pau, Barcelona, Catalonia
  - Complejo Hospitalario Virgen de las Nieves, Granada
  - Fundación Jiménez Díaz, Madrid
  - Complejo Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital la Ribera de Alzira, Valencia
  - Hospital do Meixoeiro, Vigo

REFERENCES:
- [Result] Cano A, Estevez J, Usandizaga R, Gallo JL, Guinot M, Delgado JL, Castellanos E, Moral E, Nieto C, del Prado JM, Ferrer J. The therapeutic effect of a new ultra low concentration estriol gel formulation (0.005% estriol vaginal gel) on symptoms and signs of postmenopausal vaginal atrophy: results from a pivotal phase III study. Menopause. 2012 Oct;19(10):1130-9. doi: 10.1097/gme.0b013e3182518e9a. PMID 22914208
- See also: The therapeutic effect of a new ultra low concentration estriol gel formulation (0.005% estriol vaginal gel) on symptoms and signs of postmenopausal vaginal atrophy: results from a pivotal phase III study — https://journals.lww.com/menopausejournal/Abstract/2012/10000/The_therapeutic_effect_of_a_new_ultra_low.14.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 167 patients enrolled in the study; 114 patients were randomized to the Estriol group and 53 to the placebo group.
Period: Overall Study
Arm/Group | 0.005% Estriol Group | Placebo Group
Started | 114 | 53
Completed | 105 | 48
Not Completed | 9 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Personal problems | 1 | 0
Not completed — Previous planned surgery | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population (ITT): all randomized women that received at least one dose of the study drug (Estriol gel vaginal 0.005% or placebo) after the randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.005% Estriol Group | Placebo Group | Total
Number analyzed (Participants) | 114 | 53 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 52 | 155
  >=65 years | 11 | 1 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (5.72) | 57.2 (6.70) | 56.7 (6.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 53 | 167
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 114 | 53 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Maturation Value (MV) After 12 Weeks of Treatment
Description: Maturation value (MV) is a cytologic parameter indicative of the degree of atrophy of the vaginal mucosa.
  This variable is a quantitative parameter indicative of the cytological status of the vaginal epithelium. The number of parabasal, intermediate and superficial cells was calculated from 300 consecutive cells of the samples of vaginal cytology, and the percentages of each type of cells obtained. The Maturation Value was obtained based on the following formula: 0.2 x (% parabasal) + 0.6 x (% intermediate) + 1.0 x (% superficial). The higher the value, the higher the maturation degree.
Time Frame: At week 12/Early withdrawal
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: vaginal health index
Arm/Group | 0.005% Estriol Group | Placebo Group
Number analyzed (Participants) | 114 | 53
vaginal health index | 26.9 (23.33) | 3.2 (16.48)
Statistical Analysis 1: Comparison: 0.005% Estriol Group vs Placebo Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline to Week 12 of the Vaginal pH After the 12-week Observation Period
Description: As a consequence of reduced estrogen levels, the vaginal mucosa occurs loses its rugosity, its thickness decreases, and it becomes pale and friable. The production of glycogen decreases, which determines vaginal pH alkalinization.
Time Frame: At week 12 /early withdrawal
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | 0.005% Estriol Group | Placebo Group
Number analyzed (Participants) | 114 | 53
pH units | -1.2 (1.4) | -0.4 (1.2)
Statistical Analysis 1: Comparison: 0.005% Estriol Group vs Placebo Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Number of Participants With Variation of the Individual Signs and Symptoms of Vaginal Atrophy After the 12-week Observation Period
Description: Signs and symptoms of vaginal atrophy are: vaginal dryness, pruritus or itching, burning, dyspareunia, dysuria.
  For each of these symptoms the subject indicates one the following status: present, absent, missing.
  Symptoms of vaginal atrophy were scored by the patients in a numeric scale from 0 to 3, as shown below:
  0 Absence. The symptom is not present
  1. The symptom is of mild intensity, without interfering in the patient's activity
  2. The symptom is of moderate intensity, causing obvious discomfort to the patient's
  3. The symptom is very irritating and severe in intensity
  Signs of vaginal atrophy were evaluated by the investigator and scored on a numerical scale as shown below:
  0 Absence. The symptom is not present
  1. The sign is present and is considered a mild alteration
  2. The sign is present and is considered a moderate alteration
  3. The sign is present and is considered a severe alteration
Time Frame: At baseline and at 12 weeks / early withdrawal
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 0.005% Estriol Group | Placebo Group
Number analyzed (Participants) | 114 | 53
Participants
  Vaginal dryness - Baseline - present | 114 | 53
  Vaginal dryness - Baseline - absent | 0 | 0
  Vaginal dryness - Baseline - missing | 0 | 0
  Vaginal dryness - week 12 - present: number analyzed (Participants) | 113 | 53
  Vaginal dryness - week 12 - present | 71 | 39
  Vaginal dryness - week 12 - absent: number analyzed (Participants) | 113 | 53
  Vaginal dryness - week 12 - absent | 39 | 12
  Vaginal dryness - week 12 - missing: number analyzed (Participants) | 113 | 53
  Vaginal dryness - week 12 - missing | 3 | 2
  Pruritus - Baseline - present | 55 | 29
  Pruritus - Baseline - absent | 59 | 24
  Pruritus - Baseline - missing | 0 | 0
  Pruritus - week 12 - present: number analyzed (Participants) | 113 | 53
  Pruritus - week 12 - present | 18 | 11
  Pruritus - week 12 - absent: number analyzed (Participants) | 113 | 53
  Pruritus - week 12 - absent | 92 | 40
  Pruritus - week 12 - missing: number analyzed (Participants) | 113 | 53
  Pruritus - week 12 - missing | 3 | 2
  Burning - Baseline - present | 48 | 18
  Burning - Baseline - absent | 66 | 35
  Burning - Baseline - missing | 0 | 0
  Burning - week 12 - present: number analyzed (Participants) | 113 | 53
  Burning - week 12 - present | 14 | 11
  Burning - week 12 - absent: number analyzed (Participants) | 113 | 53
  Burning - week 12 - absent | 96 | 40
  Burning - week 12 - missing: number analyzed (Participants) | 113 | 53
  Burning - week 12 - missing | 3 | 2
  Dyspareunia - Baseline - present | 101 | 48
  Dyspareunia - Baseline - absent | 11 | 5
  Dyspareunia - Baseline - missing | 2 | 0
  Dyspareunia - week 12 - present: number analyzed (Participants) | 113 | 53
  Dyspareunia - week 12 - present | 51 | 24
  Dyspareunia - week 12 - absent: number analyzed (Participants) | 113 | 53
  Dyspareunia - week 12 - absent | 56 | 25
  Dyspareunia - week 12 - missing: number analyzed (Participants) | 113 | 53
  Dyspareunia - week 12 - missing | 6 | 4
  Dysuria - Baseline - present | 27 | 14
  Dysuria - Baseline - absent | 85 | 39
  Dysuria - Baseline - missing | 2 | 0
  Dysuria - week 12 - present: number analyzed (Participants) | 113 | 53
  Dysuria - week 12 - present | 2 | 7
  Dysuria - week 12 - absent: number analyzed (Participants) | 113 | 53
  Dysuria - week 12 - absent | 108 | 44
  Dysuria - week 12 - missing: number analyzed (Participants) | 113 | 53
  Dysuria - week 12 - missing | 3 | 2

4. Secondary Outcome: Change From Baseline to Week 3 in Maturation Value (MV) After 3 Weeks of Treatment
Description: as for outcome 1
Time Frame: At week 3/ early withdrawal
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: vaginal health index
Arm/Group | 0.005% Estriol Group | Placebo Group
Number analyzed (Participants) | 114 | 53
vaginal health index | 37.9 (23.96) | 3.6 (13.15)
Statistical Analysis 1: Comparison: 0.005% Estriol Group vs Placebo Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change From Baseline to Week 3 of the Vaginal pH After the 3-week Observation Period
Description: as for outcome 2
Time Frame: At week 3 / early withdrawal
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: pH units
Arm/Group | 0.005% Estriol Group | Placebo Group
Number analyzed (Participants) | 114 | 53
pH units | -1.4 (1.4) | -0.3 (1.2)
Statistical Analysis 1: Comparison: 0.005% Estriol Group vs Placebo Group; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Variation of the Individual Signs and Symptoms of Vaginal Atrophy After the 3-week Observation Period
Description: as for outcome 3
Time Frame: At 3 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 0.005% Estriol Group | Placebo Group
Number analyzed (Participants) | 114 | 53
Participants
  Vaginal dryness - Baseline - present | 114 | 53
  Vaginal dryness - Baseline - absent | 0 | 0
  Vaginal dryness - Baseline - missing | 0 | 0
  Vaginal dryness - week 3 - present: number analyzed (Participants) | 105 | 51
  Vaginal dryness - week 3 - present | 84 | 43
  Vaginal dryness - week 3 - absent: number analyzed (Participants) | 105 | 51
  Vaginal dryness - week 3 - absent | 21 | 8
  Vaginal dryness - week 3 - missing: number analyzed (Participants) | 105 | 51
  Vaginal dryness - week 3 - missing | 0 | 0
  Pruritus - Baseline - present | 55 | 29
  Pruritus - Baseline - absent | 59 | 24
  Pruritus - Baseline - missing | 0 | 0
  Pruritus - week 3 - present: number analyzed (Participants) | 105 | 51
  Pruritus - week 3 - present | 21 | 13
  Pruritus - week 3 - absent: number analyzed (Participants) | 105 | 51
  Pruritus - week 3 - absent | 84 | 38
  Pruritus - week 3 - missing: number analyzed (Participants) | 105 | 51
  Pruritus - week 3 - missing | 0 | 0
  Burning - Baseline - present | 48 | 18
  Burning - Baseline - absent | 66 | 35
  Burning - Baseline - missing | 0 | 0
  Burning - week 3 - present: number analyzed (Participants) | 105 | 51
  Burning - week 3 - present | 22 | 11
  Burning - week 3 - absent: number analyzed (Participants) | 105 | 51
  Burning - week 3 - absent | 83 | 40
  Burning - week 3 - missing: number analyzed (Participants) | 105 | 51
  Burning - week 3 - missing | 0 | 0
  Dyspareunia - Baseline - present | 101 | 48
  Dyspareunia - Baseline - absent | 11 | 5
  Dyspareunia - Baseline - missing | 2 | 0
  Dyspareunia - week 3 - present: number analyzed (Participants) | 105 | 51
  Dyspareunia - week 3 - present | 60 | 32
  Dyspareunia - week 3 - absent: number analyzed (Participants) | 105 | 51
  Dyspareunia - week 3 - absent | 40 | 16
  Dyspareunia - week 3 - missing: number analyzed (Participants) | 105 | 51
  Dyspareunia - week 3 - missing | 5 | 3
  Dysuria - Baseline - present | 27 | 14
  Dysuria - Baseline - absent | 85 | 39
  Dysuria - Baseline - missing | 2 | 0
  Dysuria - week 3 - present: number analyzed (Participants) | 105 | 51
  Dysuria - week 3 - present | 7 | 5
  Dysuria - week 3 - absent: number analyzed (Participants) | 105 | 51
  Dysuria - week 3 - absent | 98 | 46
  Dysuria - week 3 - missing: number analyzed (Participants) | 105 | 51
  Dysuria - week 3 - missing | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study (baseline, day 1, week 3, week 8, and week 12)
Arm/Group | 0.005% Estriol Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/114 | 0/53
Other Adverse Events (participants affected / at risk) | 50/114 | 20/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.005% Estriol Group (N=114) | Placebo Group (N=53)
Crural hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.005% Estriol Group (N=114) | Placebo Group (N=53)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Synusitis (Infections and infestations) | 1 (1) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (4)
Adnexa uteri pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Bartholinitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (10) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Sensation of heavyness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disk protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 1 (1)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 2 (2)
Migraine (Nervous system disorders) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 2 (2) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Peripheral coldness (General disorders) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 4 (4)
Labile hypertension (Vascular disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Overweight (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Dysthymic disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bunion operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Wisdom teeth removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No